CLINICAL TRIAL: NCT02462564
Title: Risk Factors for Early POCD(Postoperative Cognitive Dysfunction) in the Patients With PSM(Peritoneal Surface Malignancies )Undergoing CRS(Cytoreductive Surgery) and HIPEC(Hyperthermic Intraperitoneal Chemo-therapy)
Brief Title: Risk Factors for Early POCD in the Patients With PSM Undergoing CRS-HIPEC
Status: Completed | Type: Observational
Sponsor: Wuhan University (Other)
Responsible Party: Principal Investigator, Mian Peng, Doctor, Wuhan University
Other Study IDs: HYu
Record Dates: First submitted 2015-01-30; First posted 2015-06-04 (Estimated); Last update posted 2015-08-18 (Estimated); Status verified 2015-08

CONDITIONS: Postoperative Cognitive Dysfunction
Keywords: peritoneal surface malignancies; Post operative cognitive dysfunction
MeSH Terms: conditions — Postoperative Cognitive Complications; Peritoneal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — venous blood sample
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- postoperative cognitive dysfunction: Z score>1.96
- non-postoperative cognitive dysfunction: Z score<1.96

SUMMARY:
Objectives to investigate the incidence and associated factors for early postoperative cognitive dysfunction in the patients with peritoneal surface malignancies undergoing cytoreductive surgery and hyperthermic intraperitoneal chemo-therapy(CRS-HIPEC).Methods fifty patients aged 18-65 yr were included in the research and were grouped base on the score of neuropsychological assessments which had done in the ward at 7 day before and after the surgery. The investigators monitored various indicators in the perioperative period, such as age, body weight, sex, education, duration of operation, intraoperative blood loss, cardiovascular events, amount of fluid infused per hour. Meanwhile, the concentration of serum amploid A (SAA),IL-1beta,TNF-alpha,HMGB1,S100b,cortisol and Abeta40 were measured at the various stage of the operation and 24 hours after the operation, and the differences of data between postoperative cognitive dysfunction(POCD) and Non-POCD groups were analyzed.

ELIGIBILITY:
Inclusion Criteria:

* age < 65 years or >18 years
* The patients with peritoneal surface malignancies willing to undergo the cytoreductive surgery with hyperthermic intraperitoneal chemotherapy

Exclusion Criteria:

* age < 18 years or >65 years
* several organ function severely abnormal and can not tolerate the surgery,such as suffering from severely anemia, liver and renal function disfunction, heart and cerebrovascular disease
* cognitive function was assessed by Mini-Mental State Examination (MMSE) at 1 day before operation and the score<23
* people with neurological and psychiatric disease, such as anxiety, senile dementia, stroke sequela, cerebral hemorrhage, etc
* psychiatric drug abusers
* patients reluctant to go along with the trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with peritoneal surface malignancies undergoing cytoreductive surgery and hyperthermic intraperitoneal chemo-therapy
Sampling Method: Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2014-06; Primary Completion 2015-01 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Incidence for early postoperative cognitive dysfunction in the patients with peritoneal surface malignancies undergoing cytoreductive surgery and hyperthermic intraperitoneal chemo-therapy | 12 months

SECONDARY OUTCOMES:
Risk factor for early postoperative cognitive dysfunction in the patients with peritoneal surface malignancies undergoing cytoreductive surgery and hyperthermic intraperitoneal chemo-therapy | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Mian Peng, Doctor, Principal Investigator — Zhongnan Hospital in Wuhan University
Locations (1):
- Zhongnan Hospital in Wuhan University, Wuhan, Hubei, China